CLINICAL TRIAL: NCT06175676
Title: Safety and Efficacy of Thermosensitive Hydroxybutyl Chitosan and 5-fluorouracil Assisted Endoscopic Dacryocystorhinostomy in the Treatment of Chronic Dacryocystitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Limin Zhu, Professor, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TianjinMUEH zlm
Record Dates: First submitted 2023-12-05; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Dacryocystorhinostomy; Hydroxybutyl Chitosan; Fluorouracil; Chronic Dacryocystitis
MeSH Terms: interventions — hydroxybutyl chitosan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBCS group (Experimental): Apply HBCS to the anastomosis of the nasal mucosal flap and the dacryocyst mucosal flap
  Interventions: Drug: Hydroxybutyl chitosan
- HBCS+5-FU group (Experimental): Inject 0.3ml of 5-FU solution (25mg/ml) into the nasal mucosa around the anastomosis, and apply HBCS to the anastomosis of the nasal mucosal flap and the dacryocyst mucosal flap
  Interventions: Drug: Hydroxybutyl chitosan; Drug: 5-Fluorouracil
- Gelatin Sponge group (Active Comparator): Apply gelatin sponge sheet covered with thrombin and tobramycin and dexamethasone ophthalmic ointment to the anastomosis of nasal mucosal flap and dacryocyst mucosal flap
  Interventions: Drug: Gelatin Sponge Sheet

INTERVENTIONS:
Drug: Hydroxybutyl chitosan — Apply HBCS to the anastomosis of the nasal mucosal flap and the dacryocyst mucosal flap
  Arms: HBCS group; HBCS+5-FU group
Drug: 5-Fluorouracil — Inject 0.3ml of 5-FU solution (25mg/ml) into the nasal mucosa around the anastomosis, and apply HBCS to the anastomosis of the nasal mucosal flap and the dacryocyst mucosal flap
  Arms: HBCS+5-FU group
Drug: Gelatin Sponge Sheet — Apply gelatin sponge sheet covered with thrombin and tobramycin and dexamethasone ophthalmic ointment to the anastomosis of nasal mucosal flap and dacryocyst mucosal flap
  Arms: Gelatin Sponge group

SUMMARY:
Endoscopic dacryocystorhinostomy (En-DCR) has the advantages of less surgical trauma, shorter time, less postoperative bleeding, faster recovery, and no skin scars. However, the success rate of En-DCR surgery still varies greatly between 58% and 94% , and the main reason for the failure of the surgery is the membranous closure of the anastomosis. The application of new packing materials in dacryocystorhinostomy provides some new ways to improve the success rate of En-DCR.

Hydroxybutyl chitosan (HBCS), with its non-toxicity, biocompatibility, biodegradability, antibacterial, moisturizing properties, water solubility and temperature sensitivity, is widely used in biomedicine to prevent postoperative adhesions.

5-Fluorouracil (5-FU) is an antimetabolite drug that is effective in the treatment of keloids. The application of 5-FU in glaucoma filtration surgery has demonstrated its good safety and efficacy. Studies have shown that antimetabolites as adjuvant therapy for DCR have a positive impact on improving the success rate of surgery In this study, thermosensitive hydroxybutyl chitosan will be applied to the anastomosis site of the nasal mucosal flap and the lacrimal mucosal flap, or 0.3ml of 5-fluorouracil solution (25mg/ml) was injected into the nasal mucosa around the anastomosis at the same time. The investigators would like to observe the different situations of clinical symptoms, lacrimal duct flushing, endoscopy, and bacterial flora changes in patients with chronic dacryocystitis, to compare them with the previous intraoperative packing of gelatin sponge wrapped with thrombin and Tobramycin Dexamethasone. Furthermore, the investigators intend to evaluate the safety and efficacy of HBCS and 5-FU adjuvant internal En-DCR in the treatment of chronic dacryocystitis, and provide new ideas for the adjuvant therapy of En-DCR.

DETAILED DESCRIPTION:
Endoscopic dacryocystorhinostomy (En-DCR) has the advantages of less surgical trauma, shorter time, less postoperative bleeding, faster recovery, and no skin scars. However, the success rate of En-DCR surgery still varies greatly between 58% and 94% , and the main reason for the failure of the surgery is the membranous closure of the anastomosis. The application of new packing materials in dacryocystorhinostomy provides some new ways to improve the success rate of En-DCR.

Hydroxybutyl chitosan (HBCS), with its non-toxicity, biocompatibility, biodegradability, antibacterial, moisturizing properties, water solubility and temperature sensitivity, is widely used in biomedicine to prevent postoperative adhesions.

5-Fluorouracil (5-FU) is an antimetabolite drug that is effective in the treatment of keloids. The application of 5-FU in glaucoma filtration surgery has demonstrated its good safety and efficacy. Studies have shown that antimetabolites as adjuvant therapy for DCR have a positive impact on improving the success rate of surgery In this study, thermosensitive hydroxybutyl chitosan will be applied to the anastomosis site of the nasal mucosal flap and the lacrimal mucosal flap, or 0.3ml of 5-fluorouracil solution (25mg/ml) was injected into the nasal mucosa around the anastomosis at the same time. The investigators would like to observe the different situations of clinical symptoms, lacrimal duct flushing, endoscopy, and bacterial flora changes in patients with chronic dacryocystitis, to compare them with the previous intraoperative packing of gelatin sponge wrapped with thrombin and Tobramycin Dexamethasone. Furthermore, the investigators intend to evaluate the safety and efficacy of HBCS and 5-FU adjuvant internal En-DCR in the treatment of chronic dacryocystitis, and provide new ideas for the adjuvant therapy of En-DCR.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and able to sign an informed consent form
* Age ≥18 years
* Diagnosed with chronic dacryocystitis
* Willing and able to complete all planned visits and evaluations

Exclusion Criteria:

* Those who do not meet the inclusion criteria;
* Those who are allergic to hydroxybutyl chitosan and 5-fluorouracil;
* Patients suffering from blepharitis, hordeolum, blepharitis, ectropion, keratitis, lacrimal tumor and other external eye, ocular surface and other lacrimal diseases within three months, or those who have received eye surgery;
* Patients with chronic dacryocystitis and a history of lacrimal canal placement;
* Patients with history of lacrimal duct surgery and lacrimal duct fistula;
* Patients who have used glucocorticoid sprays within three months.
* Those who have had a history of facial trauma (eyelid trauma, nasal trauma, etc.) or have undergone facial surgery within three months;
* Abnormal nasal cavity or nasal diseases (nasal polyps, nasal tumors, turbinate hypertrophy, nasal bone fracture, etc.) within three months or those who have undergone nasal surgery;
* Patients with epiphora caused by other reasons such as facial paralysis or severe eyelid laxity;
* Those who suffer from autoimmune diseases, bleeding diseases, renal insufficiency dialysis treatment and other serious systemic diseases
* Patients with blisters or herpes zoster;
* Those with more serious skin diseases such as acne, rosacea or scar constitution;
* According to the investigator's judgment, it may interfere with Test results or medical history, personal history and allergy history that increase the risk of patients;
* Those who have participated in clinical trials of other drugs within the last 3 months;
* Those who cannot be followed up regularly or who cannot cooperate with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms | six moths
  postoperative comfort and bleeding, and epiphora using score sheets

SECONDARY OUTCOMES:
Lacrimal duct flushing | six moths
  Check for patency of the lacrimal drainage

OTHER OUTCOMES:
Endoscopic examination | six moths
  anastomotic areas(the lengths of the long and short axes), scarring and adhesions, and granulation
Bacterial flora changes | two moths
  conjunctival sac, nasal mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Li min, Study Director — Tianjin medical university eye hosipital
Locations (1):
- Limin Zhu, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT06175676/Prot_SAP_ICF_000.pdf